CLINICAL TRIAL: NCT05957809
Title: The Effects of Structured Exercise Training on Disease Course in Newly Diagnosed Multiple Sclerosis
Brief Title: Structured Exercise Training in Newly Diagnosed Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Feray Güngör, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023/68
Record Dates: First submitted 2023-06-20; First posted 2023-07-24 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; newly diagnosis; exercise; postural sway; cognition
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1. Structured exercise group (Experimental): This group will receive structured exercise training with 60-75 minute sessions per day, 2 days a week, for 8 weeks.
  Interventions: Other: Structured exercise training
- 2. Control group (No Intervention): This group will be assessed at the beginning, 8. and 24. weeks.

INTERVENTIONS:
Other: Structured exercise training — This group will receive structured exercise training with 60-75 minute sessions per day, 2 days a week, for 8 weeks. • Warm-up program - 10 minutes
  * Strength training on unstable surfaces - 25-30 minutes
  * High repetition muscular endurance training - 25-30 minutes
  * Cool-down program - 10 minutes
  Arms: 1. Structured exercise group

SUMMARY:
the effectiveness of structured exercise training will be investigated for individuals with MS who are newly diagnosed and have no clinical problems. Individuals with MS included in the study will be randomly divided into two groups a Structured Exercise Group (SEG) and a Control Group (CG). In order to compare baseline and follow-up data, the Healthy Group (HG) will be taken and all three groups will be evaluated initially, 8. weeks and 24. weeks with primary and secondary outcome measurements. SEG, CG, and HG will be evaluated initially for postural sway, muscle strength, mobility, dexterity, cognitive function, trunk strength-endurance, and fatigue. Afterward, SEG will receive structured exercise training consisting of clinically supervised aerobic exercise and resistance training on unstable surfaces for 8 weeks, 2 days a week, with a minimum session duration of 60 minutes. Stretching and mobility exercises will be added to warm up and cool down before and after the program. CG will be on the waiting list during this process. At the end of 8 weeks, both groups will be reassessed with their initial assessment. After the 8-week program, the SEG physical activity recommendation will be given and the KG group will continue on the waiting list, and a follow-up evaluation will be made in the 24th week. This study will allow the comparison of newly diagnosed individuals with MS who do not have any physical or cognitive effects on neurological examination and healthy controls with objective and detailed evaluations, and will also reveal the evidence on the effects of planned structured exercises specific to individuals with newly diagnosed MS. During the 24-week follow-up period, the change in the clinical status of individuals with MS who received or did not receive any exercise training can be interpreted.

DETAILED DESCRIPTION:
According to the data of the World Multiple Sclerosis (MS) atlas, the incidence of MS in our country is 51-100/100.000 and it is estimated that there are over 70.000 individuals with MS. MS continues to be the most common cause of non-traumatic neurological disability in young adults with its increasing prevalence in our country as well as all over the world. The most common problems seen in MS are deterioration of balance and postural control, decrease in muscle strength, gait problems, and cognitive and emotional functions. These effects become more visible in the later stages of the disease, but a limited number of studies reveal that there is an insidious progression from the early period. The topographical model of MS suggests that the burden of disease below the threshold is compensated by functional reserve, presents no physical problems, and symptoms become evident once the clinical threshold is crossed. Furthermore, the evidence suggests that disease activity may be continued even during the relapse-remitting phase of the disease course, highlighting the need for the use of sensitive outcome measures that can detect early disorders. Therefore, the involvement in individuals with newly diagnosed MS is ignored because it is not reflected in activities of daily living, is compensated by functional reserve because it is below the threshold value, and cannot be detected in the non-objective clinical neurological examination. Rehabilitation approaches for individuals with newly diagnosed MS are needed in order to benefit from the protective effects of exercise and to prevent the effects from progressing. Therefore, within the scope of our proposed project, the effectiveness of structured exercise training will be investigated for individuals with MS who are newly diagnosed and have no clinical problems. Individuals with MS included in the study will be randomly divided into two groups a Structured Exercise Group (SEG) and a Control Group (CG). In order to compare baseline and follow-up data, the Healthy Group (HG) will be taken and all three groups will be evaluated initially, 8. weeks and 24. weeks with primary and secondary outcome measurements. SEG, CG, and HG will be evaluated initially for postural sway, muscle strength, mobility, dexterity, cognitive function, trunk strength-endurance, and fatigue. Afterward, SEG will receive structured exercise training consisting of clinically supervised aerobic exercise and resistance training on unstable surfaces for 8 weeks, 2 days a week, with a minimum session duration of 60 minutes. Stretching and mobility exercises will be added to warm up and cool down before and after the program. CG will be on the waiting list during this process. At the end of 8 weeks, both groups will be reassessed with their initial assessment. After the 8-week program, the SEG physical activity recommendation will be given and the KG group will continue on the waiting list, and a follow-up evaluation will be made in the 24th week. This study will allow the comparison of newly diagnosed individuals with MS who do not have any physical or cognitive effects on neurological examination and healthy controls with objective and detailed evaluations, and will also reveal the evidence on the effects of planned structured exercises specific to individuals with newly diagnosed MS. During the 24-week follow-up period, the change in the clinical status of individuals with MS who received or did not receive any exercise training can be interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with MS according to McDonald diagnostic criteria
* EDSS below 2.5
* Diagnosis period less than 1 year
* Being between the ages of 18-45
* Volunteering to participate in the study

Exclusion Criteria:

* Apart from the MS diagnosis, orthopedic, neurological, psychological, etc., which will affect the evaluation results. have diseases
* Regular exercise and doing sports
* Being involved in another rehabilitation program
* Being pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Clinical Test of Sensory Integration of Balance Test | 24 weeks
  Postural sway in "open eyes-firm surface, closed eyes-firm surface, open eyes-foam surface, closed eyes-foam surface" conditions will be evaluated with the Clinical Test of Sensory Integration of Balance.
Postural Stability Test | 24 weeks
  Anterior-posterior, mediolateral and overall sway will be evaluated with the Postural Stability Test in Biodex Balance System.
Balance Error Scoring System Test | 24 weeks
  Postural sway in tandem position and feet together position will be evaluated with Balance Error Scoring System in Biodex Balance System.
Muscle strength | 24 weeks
  Quadriceps, hamstring, ankle dorsi and plantar flexors muscle strength will be assessed with Hand Held Dynamometer.

SECONDARY OUTCOMES:
2 Minute Walk Test | Baseline, 8th and 24th weeks
  It will be used to evaluate walking speed.
Timed 25 Foot Walk Test | Baseline, 8th and 24th weeks
  It will be used to evaluate walking distance.
Brief International Cognitive Assessment for MS (BICAMS) | Baseline, 8th and 24th weeks
  BICAMS will be used to evaluate cognitive functions.
Curl-up | Baseline, 8th and 24th weeks
  It will be used to evaluate trunk flexor muscle strength. While the hips and knees are in 90º flexion position and the feet are fixed by the therapist, the individuals will be asked to flex their trunk and the number of repetitions done for 30 seconds will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Feray Güngör, Istanbul, Turkey (Türkiye)